CLINICAL TRIAL: NCT02567994
Title: Efficacy and Safety of Teneligliptin Versus Sitagliptin as add-on Therapy to Metformin Plus Glimepiride in T2DM Patinets With Inadequate Glycemic Control
Brief Title: Tenelia Triple Combination Study
Acronym: TETRIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP_C303
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teneligliptin (Experimental): 20mg qd
  Interventions: Drug: Teneligliptin
- Sitagliptin (Active Comparator): 100mg qd
  Interventions: Drug: Teneligliptin

INTERVENTIONS:
Drug: Teneligliptin — Subjects will visit the center on Week 4, 12 and 24 during the entire 24-week treatment period. Total study duration will be approximately 28weeks and the subjects will be to practice exercise/diet control together.

SUMMARY:
After a screening, a 2-week, single-blind placebo run-in, 200 patients will be randomized in a 1 : 1 ratio to the addition of either once-daily Teneligliptin 20mg or sitagliptin 100mg to ongoing stable doses of glimepiride in combination with metformin for 24 weeks.

DETAILED DESCRIPTION:
Subjects will visit the centers on Week 4, 12 and 24 during the entire 24-week treatment period. Total study duration will be approximately 28weeks and the subjects will be to practice exercise/diet control together.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Type 2 Diabetes Mellitus
2. Adults aged ≥ 19 years old
3. Patients with HbA1c 7%~11% at Screening and Run-in visit

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change of HbAlc from baseline at Week 24 | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes